CLINICAL TRIAL: NCT04005118
Title: Human Intestinal Microbiome and Surgical Outcomes in Patients Undergoing Colorectal Cancer Surgery
Acronym: Microbiota
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190088
Record Dates: First submitted 2019-03-15; First posted 2019-07-02 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-05

CONDITIONS: Adenocarcinoma of the Colon; Adenocarcinoma of the Rectum
Keywords: Intestinal microbiome; colorectal cancer; mechanical bowel preparation; postoperative complications; anastomotic leakage
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Colorectal Neoplasms; Postoperative Complications; Anastomotic Leak

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 3 different microbiome samples will be taken from all patients. Two fresh fecal samples for detection of luminal microbiota (LM) and fecal water preparation: a) a day before the surgery before Mechanic Bowel Preparation (MBP) and/or antibiotics (ABT) (LM1), b) postoperatively after first bowel movement (LM2). One sample will be taken intra-operatively from the stapled resection lines of circular stapler used for forming a colorectal anastomosis, to detect the Mucosal Associated Microbiota (MAM) and to perform immunohistochemistry staining for detection of HACE1 expression.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- preoperative preparation on microbiome composition: Mechanical Bowel Preparation + oral antibiotics group: receiving mechanical bowel preparation only MBP will be prepared with 4 liters of Polyethylene glycol (PEG) solution to be started 24 hours before the planned surgery. 500mg of Metronidazole will be administrated 3 times one day before the surgery at 2 pm, 3 pm and 10 pm.

SUMMARY:
Intro: Recent studies on colorectal cancer surgery have been focusing on the role of intestinal microbiome on surgical outcomes. Standard perioperative cares, like mechanic bowel preparation (MBP), administration of antibiotics (ABT) and surgery-related stress and injury influence the microbiome composition and possibly induce a shift toward a microbiome dysbiotic state, which predisposes to complicated postoperative course. Microbiome composition changes and enhanced virulence factors may increase the risk of postoperative complications, such as anastomotic leakage (AL), surgical site infection (SSI), and postoperative ileus (PI), which are known to impact on patient's overall survival and cancer recurrence.

Objective: The primary objective is to investigate if a significant association might exist between the microbiome composition and the occurrence of postoperative complications at 90 days.

Methods: 3 different microbiome samples will be taken from all patients. Two fresh fecal samples for detection of LM and fecal water preparation: a) a day before the surgery before MBP and/or ABT (LM1), b) postoperatively after first bowel movement (LM2). One sample will be taken intra-operatively from the stapled resection lines of circular stapler used for forming a colorectal anastomosis, to detect the MAM and to perform immunohistochemistry staining for detection of HACE1 expression.

DNA analysis will be performed for all samples. IHC will be performed for detecting HACE1 expression in the tumor and colorectal anastomosis tissues using anti-HACE1 antibodies. .

For proliferation assessment, human colon carcinoma cell lines HT29 will be plated in monolayers and scratched with a single scratch. Monolayers will be incubated for 24 hours with fecal water from patients with surgical complications and matched control patients without complications.

Descriptive statistics will be performed to describe the study population. This project aim to describe microbiome composition and its impact on postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥ 18 years old
* With histologically confirmed rectal or left colon adenocarcinoma by biopsy material from colonoscopy
* Having elective colorectal surgery after standardized bowel preparation
* Affiliated to a social security system
* Signature of informed consent

Exclusion Criteria:

* Major surgery 30 days before scheduled colorectal surgery
* Administration of systemic antibiotic therapy within 30 days prior to planned colorectal surgery
* Presenting a contraindication to elective colorectal surgery
* Patient protected by law
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with rectal or left colon adenocarcinoma
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-05-28 (Actual); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
Rate of anastomotic leakage | 90 days after surgery
  detected by imaging techiques (CT scan or MRI)
Rate of surgical site infection | 90 days after surgery
  1)superficial and deep infection:clinical observation of purulent discharge from the wound and/or bacterial staining from the wound 2)organ or deep space infection: imaging techniques (CT, MRI, USS)
Rate of prolonged postoperative ileuss | 90 days after surgery
  detected by clinical observation of the first bowel movement after the surgery

SECONDARY OUTCOMES:
microbiome composition | 3 months after study start date
  The composition of luminal microbiome and mucosal-associated microbiome will be studied by DNA analyses from fresh fecal samples and surgical anastomosis material, accordingly
microbiome composition | 6 months after study start date
  The composition of luminal microbiome and mucosal-associated microbiome will be studied by DNA analyses from fresh fecal samples and surgical anastomosis material, accordingly
impact of microbiome composition on length of hospitalization | at the time of patient's discharge of the hospital
  length of hospitalization will be detected and analyzed in association with microbiome composition
Correlation between detected bacterial OTUs (Operation Taxonomic Units) and the event of reintervention | 90 days after surgery
  In the patient group with the event of reintervention, an abundance of specific OTUs will be analysed in compare with patients with no event of reintervention.
impact of microbiome metabolites on intestinal epithelial cell proliferation and wound healing | 6 months after study start date
  Monolayers of human colon cancer cell lines HT29 will be incubated for 24 hours with fecal water from patients with surgical complications and matched control patients without complications.
  Proliferation will be calculated in two manners: 1) The time of the closure of the scratch defect will be evaluated and compared in the two group., 2)Proliferation rate will be analyzed by immunohistochemistry marker Ki 67, expression of Ki 67 will be evaluated in cells at the borders of the scratch defect
Expression intensity in cytoplasm of protein ligase HACE1 in tumoral and non-tumoral tissues | 6 months after study start date
  Immunohistochemistry with anti-HACE1 antibodies will be used to detect expression levels in tumoral (colorectal cancer) and non-tumoral (anastomotic sample) tissues. In a case of decreased expression, tissues will be analyzed by methylation PCR to detect an aberrant methylation of HACE1 and its hypermethylation
Expression intensity in cytoplasm of protein ligase HACE1 in tumoral and non-tumoral tissues | 3 months after study start date
  Immunohistochemistry with anti-HACE1 antibodies will be used to detect expression levels in tumoral (colorectal cancer) and non-tumoral (anastomotic sample) tissues. In a case of decreased expression, tissues will be analyzed by methylation PCR to detect an aberrant methylation of HACE1 and its hypermethylation

CONTACTS AND LOCATIONS:
Overall Officials: Lelde Lauka, PHD, Principal Investigator — APHP
Locations (1):
- Dr Lelde Lauka, Créteil, France

IPD SHARING:
Plan to Share IPD: No
DATAS ARE OWN BY ASSISTANCE PUBLIQUE - HOPITAUX DE PARIS, PLEASE CONTACT SPONSOR FOR FURTHER INFORMATION